CLINICAL TRIAL: NCT00613743
Title: Effect of Topical Morphine (Mouthwash) on Oral Pain Due to Chemo- and/or Radiotherapy Induced Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Pautex Sophie, university hospital geneva
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-165/psy06-033
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2008-01

CONDITIONS: Cancer; Mucositis
MeSH Terms: conditions — Neoplasms; Mucositis | interventions — Mouthwashes; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): D1-D3 receive placebo
  Interventions: Drug: placebo
- 2 (Active Comparator): receive D1 D3 morphine
  Interventions: Drug: mouth wash with morphine

INTERVENTIONS:
Drug: mouth wash with morphine — morphine solution 0.2% concentration; 15ml per unit mouthwash 6 time à day
  Arms: 2
Drug: placebo — placebo solution Quinine diHCl 0.3% at 50 mg/15 ml mouthwash 6 time/day
  Arms: 1

SUMMARY:
Introduction:

Oral pain due to mucosal lesion is quite frequent in oncology, geriatric as well as palliative care settings. The oncology patient is mainly suffering from radio- and/or chemotherapy induced oral mucositis. The incidence of oral mucositis in oncology patients ranges from 15-40% in those receiving stomatotoxic chemotherapy or radiotherapy. The degree of mucositis is variable, but the associated pain is frequent and well documented. Nowadays, basic oral care protocols are the mainstay of preventing or reducing mucositis pain. Pain is mainly managed by systemically administered analgesia. The only pioneer work in the field of radio-or chemotherapy induced mucositis treatment with topical opioids has been done by Cerchietti in two pilot studies: one compared "magic" mouthwash (lidocaine, diphenhydramine, magnesium aluminium hydroxide) with morphine mouthwash in a randomized trial; the other compared 1%o and 2% morphine solutions in an open trial. The results showed a significant decrease in the duration of pain, the intensity as well as a decrease the need for systemic analgesia in the group with morphine mouthwash. No systemic clinically relevant adverse effects were noted.

Hypothesis:

Mouthwashes with a morphine containing solution decrease oral pain substantially, while not causing the side effects seen in systemic administration of narcotic analgesics.

Method:

A randomised double-blind cross-over study to evaluate the effect of topical oral application of a 0.2% morphine solution in patients suffering from radio- and/or chemotherapy induced oral mucositis. 60 patients will be included. Randomly assigned to either the morphine solution or a placebo mouthwash, they receive the first three days one of the solutions and then are switched over to the other treatment for three more days. General basic oral care is offered to all of the patients. Efficacy of treatment will be measured with a self-assessment pain scale. Doses of systemic opioids and other symptoms (appetite, dysphagia) will also be measured. If patient's don't receive systemic opioids, serum concentrations of morphine will be measured.

DETAILED DESCRIPTION:
randomised double-blind cross-over study to evaluate the effect of topical oral application of a 0.2% morphine solution in patients suffering from radio- and/or chemotherapy induced oral mucositis. 60 patients will be included. Randomly assigned to either the morphine solution or a placebo mouthwash, they receive the first three days one of the solutions and then are switched over to the other treatment for three more days. General basic oral care is offered to all of the patients. Efficacy of treatment will be measured with a self-assessment pain scale. Doses of systemic opioids and other symptoms (appetite, dysphagia) will also be measured. If patient's don't receive systemic opioids, serum concentrations of morphine will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalised patients, or ambulatory patients that have daily radiotherapy in HUG
* No risk of swallowing the mouth wash solution (determined before inclusion by a recovery of more than 90% of the 15ml of water solution used for testing)
* Treatment with chemo- and/or radiotherapy causing oral mucositis
* Oral pain associated with mucosal injury (WHO grading of mucositis >= 2)
* Cognition: Mini Mental Status Examination of at least 28/30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
difference of pain alleviation in the two branches one hour after mouthwash and as well as the duration of pain relief. | 1 year

SECONDARY OUTCOMES:
the requirement of supplementary systemic analgesics | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Pautex, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Collonge-bellerive, Switzerland